CLINICAL TRIAL: NCT05750667
Title: Leveraging Behavioral Economics to Equitably Implement Cascade Screening in Individuals With Familial Hypercholesterolemia in Partnership With the FH Foundation (R33 Phase)
Brief Title: Penn Family Screening for Familial Hypercholesterolemia
Acronym: NHLBI-R33
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: University of Pennsylvania (Other); Family Heart Foundation (Unknown)
Responsible Party: Principal Investigator, Rinad Beidas, Ralph Seal Paffenbarger Professor and Chair, Department of Medical Social Sciences, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SP0078729
Record Dates: First submitted 2023-02-15; First posted 2023-03-02 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Familial Hypercholesterolemia
Keywords: implementation science; behavioral economics; equity; cascade screening
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Intervention Model Description: Probands will be randomized to one of the two active implementation strategy arms (Penn Medicine, Family Heart Foundation; n=220 each) or usual care (n=360).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Penn Medicine (health system)-mediated (Experimental): Probands receive automated text messages and/or emails through the Way to Health (WTH) platform containing information about FH and cascade screening from Penn Medicine, and a request to identify first-degree biological relatives. Probands choose whether to contact relatives themselves or share contact information so that automated text messages and/or emails can be sent by Penn Medicine to relatives directly via WTH. If probands opt to contact relatives themselves (self-contact), they receive tips on how to do this effectively. If probands opt for Penn Medicine to contact their relatives (direct contact), relatives receive information via WTH about FH and instructions for screening. All relatives (regardless of whether they were contacted via self-contact and direct contact) will be offered FH screening at no cost. If a proband's initial choice of outreach is not successful, they will have the option of initiating the alternate outreach approach (direct or self-contact).
  Interventions: Behavioral: Cascade screening
- Family Heart Foundation-mediated (Experimental): After using WTH to conduct an identity screen and giving probands an option to opt-out of having their information shared with Family Heart Foundation (FHF), FHF reaches out directly to probands via an FHF-employed navigator. During an initial call, the navigator introduces the proband to navigation services, conducts a social history, and initiates a plan for contacting relatives. Probands choose whether to contact relatives themselves (self-contact) or have FHF contact relatives directly (direct contact). Those who choose self-contact receive personalized coaching to address barriers and concerns. For direct contact relatives, FHF will call these relatives directly. All relatives (regardless of whether they were contacted via self-contact and direct contact) will be offered FH screening at no cost. If a proband's initial choice of outreach is not successful, they will have the option of initiating the alternate outreach approach (direct or self-contact).
  Interventions: Behavioral: Cascade screening
- Usual Care (No Intervention): Probands randomized to this arm will not receive any contact from the research team or Family Heart Foundation regarding cascade screening (i.e., no intervention).

INTERVENTIONS:
Behavioral: Cascade screening — FH is a genetic condition that causes high LDL cholesterol starting at birth. When one individual with FH is diagnosed, it is important that biological family members are also screened, since there is a 50% chance that each first-degree relative will have also inherited FH. More distant relatives may also have inherited FH. This evidence-based process is known as cascade screening.
  Arms: Family Heart Foundation-mediated; Penn Medicine (health system)-mediated

SUMMARY:
The goal of this clinical trial is to test two implementation strategies (automated health system [Penn Medicine]-mediated strategy vs. Family Heart Foundation-mediated strategy using a patient navigator) versus usual care to promote family cascade screening for familial hypercholesterolemia (FH) in Penn Medicine patients diagnosed with FH ("probands"). The main questions this study aims to answer are: (1) evaluating the effect of the three approaches on reach (proportion of probands who have at least one family member who completes screening), number of family members screened, number of family members diagnosed with FH, and proband LDL-C levels; and (2) identifying implementation strategy mechanisms focusing on health equity using mixed methods and oversampling populations that experience disparities. Participants (probands) in the active arms (health system [Penn Medicine]-mediated, Family Heart Foundation-mediated) will receive messaging that provides education about FH and provides instructions for participating in family cascade screening. A subset of probands will be invited to complete a qualitative interview about their experience receiving the implementation strategy. The research team will compare the active arms to Penn Medicine usual care for cascade screening to evaluate whether the active arms are more effective at promoting cascade screening than usual care.

DETAILED DESCRIPTION:
This project leverages Penn Medicine's and the investigative team's longstanding partnership with the Family Heart Foundation (FHF), a nonprofit research and advocacy organization, to test two promising approaches to implementing cascade screening. The study will test two patient-facing implementation strategies to increase reach of cascade screening with FH probands within Penn Medicine. This pragmatic randomized controlled trial (RCT) will test (a) a health system (Penn Medicine)-mediated strategy using automated text messages and emails, (b) an FHF-mediated strategy delivered by a navigator, and (c) the "usual care" approach. Both active strategies use centralized direct contact to relatives and behavioral economics. Specifically, we will conduct a 3-arm hybrid type III effectiveness-implementation RCT.

Aim 1: Compare the effect of the three arms on effectiveness and implementation outcomes.

* Reach (primary outcome): proportion of probands who have at least one family member who completes screening
* Absolute number of family members screened
* Absolute number of family members with a new FH diagnosis
* Proband LDL-C levels 12 months post-randomization

Aim 2: Use mixed methods to identify implementation strategy mechanisms with a focus on health equity. In Aim 2a, the researchers will conduct qualitative interviews to understand proband perspectives on mechanisms of the implementation strategies using the Consolidated Framework for Implementation Research, oversampling for populations at risk for disparities. In Aim 2b, the researchers will explore disparities quantitatively by evaluating differential strategy effectiveness by race/ethnicity and gender; and descriptively explore differential strategy effectiveness by income and medical mistrust.

ELIGIBILITY:
Inclusion Criteria (probands):

* Adults aged 18 years and older with clinically diagnosed FH who are treated within the Penn Medicine system
* Have contact information for at least one living, first-degree biological relative
* Have a cell phone with texting capabilities and/or access to email

Exclusion Criteria (probands):

* People under age 18
* Do not have contact information for at least one living, first-degree biological relative
* Do not have a cell phone with texting capabilities nor access to email

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2023-01-24 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Reach | Collected from proband randomization date through six months post-randomization
  Reach is defined as the proportion of probands who have at least one family member who completes screening (via a lipid panel or an FH genetic test) within 6 months of proband randomization. To mimic real world settings, we will allow family members to select how they would like to complete their screening from a range of mechanisms: sharing results from a recent lipid panel, requesting a lipid panel from their primary care provider, or having the study clinician order a lipid panel via LabCorp, a nationwide lab testing company.

SECONDARY OUTCOMES:
Absolute number of family members who are screened for FH as a result of cascade screening | Collected from proband randomization date to six months post-randomization
  Absolute number of family members who are screened for FH as a result of cascade screening within 6 months of proband enrollment will be obtained through several complementary approaches: 1) self-report from the proband or from the family member; 2) confirmation of lipid testing by the study; 3) direct receipt of blood lipid panel testing from the lab when ordered by the study clinician.
Absolute number of family members who are newly diagnosed with FH as a result of cascade screening | Collected from proband randomization date to six months post-randomization
  Absolute number of family members who are newly diagnosed with FH as a result of cascade screening within 6 months of proband enrollment will be obtained through several complementary approaches: 1) self-report from the proband or from the family member; 2) confirmation of genetic testing by the study; 3) direct receipt of genetic testing from the lab when ordered by the study clinician.
LDL-C in probands | One-time collection at 12 months post-randomization
  Proband LDL-C will be collected via lipid panel results obtained through two complementary approaches: 1) self-report from the proband; or 2) direct receipt of blood lipid panel testing from the lab when ordered by the study clinician.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Perelman School of Medicine, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Johnson C, Chen J, McGowan MP, Tricou E, Card M, Pettit AR, Klaiman T, Rader DJ, Volpp KG, Beidas RS. Family cascade screening for equitable identification of familial hypercholesterolemia: study protocol for a hybrid effectiveness-implementation type III randomized controlled trial. Implement Sci. 2024 Apr 9;19(1):30. doi: 10.1186/s13012-024-01355-x. PMID 38594685

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT05750667/Prot_SAP_000.pdf